CLINICAL TRIAL: NCT01115647
Title: Treating Moderate Malnutrition in 6-24 Months Old Children: Acceptability, Efficacy and Cost-effectiveness of a Local Soy-based RUTF vs. Enhanced Corn Soy Blend vs. Child-centered Counselling
Brief Title: Treating Moderate Malnutrition in 6-24 Months Old Children
Acronym: LUCOMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Tropical Medicine, Belgium (Other)
Collaborators: Institut de Recherche en Sciences de la Sante, Burkina Faso (Other Government); Ministry of Health, Burkina Faso (Other Government); University Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ITMH0110
Record Dates: First submitted 2010-04-29; First posted 2010-05-04 (Estimated); Last update posted 2011-11-22 (Estimated); Status verified 2011-11

CONDITIONS: Moderate Acute Malnutrition
Keywords: Malnutrition; Nutritional intervention; Behavioural intervention; Burkina Faso; Cluster randomize trial
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Ready-to-Use Therapeutic Foood (RUSF) (Experimental): Caretakers will receive weekly RUSF, 350g, and will be advised to feed it(50 g d-1 or 3 tablespoons/day) in one meal or on demand. These are pre-defined quantities. However, minimum quantities required for a timely (≤15 days) recovery from moderate malnutrition will be determined during the pilot phase.
  Besides supplementary food, parents will be provided with the usual nutrition counsels prevailing currently in the health services.Children will be home-visited once a week by assessors for anthropometry, 24-hours recall of dietary and breastfeeding intake, and morbidity signs. Feeding practices will be assessed, and the changes between baseline and intervention periods evaluated. Compliance will be evaluated by interviewing family members.
  Interventions: Dietary Supplement: Ready-to-Use Therapeutic Food (RUTF)
- CSB++ (Active Comparator): Caretakers will receive weekly CSB++ (450g) rations. Parents will be advised to feed the CSB++ (65g d-1 diluted in 370 g water) in one meal or on demand. These are pre-defined quantities. However, minimum quantities of CSB++ required for a timely (≤15 days) recovery from moderate malnutrition in the area will be determined during the pilot phase. Besides supplementary foods, parents will be provided with the usual nutrition counsels prevailing currently in the health services, i.e. to keep on breastfeeding, to increase diet diversity and to feed frequent snacks.
  Feeding practices will be also assessed, and the changes between baseline and intervention periods evaluated. Compliance will be evaluated by interviewing family members.
  Interventions: Dietary Supplement: CBS++
- Children Centered Counseling (CCC) (Active Comparator): The counsellor will spend 1 hour daily (during the 3 first days and then weekly) within the household for identifying enhancing and blocking factors and adapt consequently the treatment strategies in agreement with the caretakers.
  As in the other study arms, children will be home-visited once a week by assessors for anthropometry, 24-hours recall of dietary and breastfeeding intake, and morbidity signs. Feeding practices will be also assessed in each arm, and the changes between baseline and intervention periods evaluated. Compliance will be evaluated by interviewing family members.There will be no dietary supplements intervention, outside normal practices in Burkina.
  Interventions: Behavioral: CCC

INTERVENTIONS:
Dietary Supplement: Ready-to-Use Therapeutic Food (RUTF) — A Ready-to-Use Therapeutic Food (RUTF), locally produced in Burkina Faso. The RUSF will be nutritionally characterized by chemical analysis (macronutrients, amino acids, vitamins A, C, D, E, B12, thiamin, riboflavin, niacin, calcium, iron, zinc, copper, selenium) and will be analyzed for macronutrients and energy density. All analysis methods are either based on the Official Methods of Analysis of AOAC International or in-house validated analytical methods. The pilot production phase and Hazard Analysis of Critical Control Points (HACCP) risk inventory of the production process will be performed by a food technologist from the Department of Food safety and Food quality, Ghent University.
  Arms: Ready-to-Use Therapeutic Foood (RUSF)
Dietary Supplement: CBS++ — CSB is a low-cost combination of a cereal and a legume sometimes fortified with micronutrients. However, it presents shortcomings such as too many anti-nutrients, suboptimal micronutrient content, high bulk and viscosity. The World Food Program has recently proposed an enhanced CSB, named CSB++, which is prepared from heat treated maize and de-hulled soya beans, sugar, dried skim milk, refined soya bean oil, vitamins and minerals.
  Arms: CSB++
Behavioral: CCC — Child-Centred dietary Counselling (CCC). Although educational/behavioral interventions can be effective to improve child growth, there is little evidence of their effectiveness for MAM. Moreover, evidence from Africa is inexistent. Currently, the main management of MAM consists of giving nutritional advice to the caretakers, but mothers of MAM children are given the same general dietary advice as mothers of well-nourished children. A more efficient, child-centred approach is therefore proposed, by adapting the counselling to the needs of the family, developing a more child-centred approach, by providing operational recommendations for MAM children and providing an adequate follow-up post-treatment.
  Arms: Children Centered Counseling (CCC)

SUMMARY:
Child malnutrition is intimately associated to poverty and may be due to sub-optimal feeding behaviours, food insecurity at household level, or a combination of both. Acute malnutrition is a major contributor to under-5 mortality and morbidity in developing countries. While clinical guidelines for severe acute malnutrition (SAM) have been available for a decade, research on the management of moderate acute malnutrition (MAM) has lagged behind. Nonetheless, MAM is much more incident than SAM, it increases mortality risk by itself and requires special nutritional treatment. This study is thus meant to address this major gap, by testing the relative feasibility, effectiveness and cost-effectiveness of three innovative strategies for treating children with MAM aged 6-24 months : a locally produced Ready-to-Use Therapeutic Food (RUTF), a corn/soy blended flour (CSB++)provided by the World Food Program, and a specific and context-appropriate child-centred counselling.

The evaluation will be carried out as a cluster-randomized trial in the Houndé district, Burkina Faso, where 18 rural health centres will be randomly allocated to RUSF or CSB or CCC for treating MAM.

DETAILED DESCRIPTION:
Child malnutrition is intimately associated to poverty and may be due to sub-optimal feeding behaviours, food insecurity at household level, or a combination of both. Acute malnutrition is a major contributor to under-5 mortality and morbidity in low and middle income countries. Clinical guidelines for the management of severe acute malnutrition (SAM) have been available for a decade and have yielded excellent results. However, the corresponding research on the management of moderate acute malnutrition (MAM) has lagged behind, even if MAM is much more incident than SAM, increases mortality risk on its own and requires special nutritional treatment. Currently, the main management of MAM, in Burkina Faso as in most African countries, consists of giving nutritional advice to the caretakers, but mothers of MAM children are usually given the same general dietary advice as mothers of well-nourished children. A more efficient, child-centred approach must be developed, by adapting the counselling to the needs of the family, by developing a more child-centred approach, by providing operational recommendations for MAM children, and by providing an adequate follow-up post-treatment.

This study is thus meant to address this major gap, by testing the relative feasibility, effectiveness and cost-effectiveness of three innovative strategies for treating children with MAM: a locally produced Ready-to-Use Therapeutic Food (RUTF), an enhanced corn/soy blended flour (CSB++)provided by the World Food Program, and a specific and context-appropriate child-centred counselling.

The evaluation will be based on a cluster-randomized trial carried out in the Houndé district, Burkina Faso. Eighteen rural health centres and the population living in their catchment area will be randomly allocated to RUSF or CSB or CCC for treating MAM. Only children aged 6-24 months will be included as the risk of acute malnutrition is high and more amenable to interventions in this age range. Overall, 2088 children with MAM will participate. In each study arm, children will be home-visited once a week by assessors for anthropometry, 24-hours recall of dietary and breastfeeding intake, and morbidity signs. Feeding practices will be also assessed in each arm, and the changes between baseline and intervention periods evaluated. Compliance will be evaluated by interviewing family members.

ELIGIBILITY:
Inclusion Criteria:

* living in the catchment area of one of the 18 health centres participating in this cluster randomized trial
* 6-24 months of age
* -3≤ weight for height z score <-2 without edema
* No major clinical complications
* Showing appetite

Exclusion Criteria:

* Weight-for-Height Z-score <-3 and/or the presence of bilateral
* Presence of bilateral pitting oedema
* Not showing appetite

Ages: 6 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2088 (Actual)
Dates: Start 2010-07; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Recovery rate | One month (average)
  Weight-for-Height Z-score≥-1 SD
Morbidity rate | One month (average)
  ARI, diarrhoea, anaemia and malaria incidence. Morbidity will be assessed every week by a locally pre-tested standardized questionnaire
Cost-effectiveness | Twelve months
  The net differential costs and key outcomes for each intervention will be used to calculate the incremental cost-effectiveness ratios, i.e. the incremental costs divided by the incremental benefits. Specific cost-utility analysis will be performed to disentangle costs of a routine program including the intervention elements from those incurred from the research activities of the project.

SECONDARY OUTCOMES:
Time to recovery | One month (average)
Relapse rate | Up to three months (average)
  Patients representing inclusion criteria within 3 months following discharge
Failure rate | 8 weeks
  Patients not gaining weight after 2 weeks or with a Weight-for-Height Z-score<-1 SD after 8 weeks
Default rate | 2 weeks
  Patient absent or refusing food during 2 consecutive weeks
Satisfaction of parents and acceptability | Three months (average)
  Survey to be conducted with households
Diet replacement & Intra-household dispatching of the food supplements | Three months (average)
  Assessment with households
Retinol & soluble serum transferrin receptors (Iron markers) | Three months (average)
  Retinol & soluble serum transferrin receptors (Iron markers)

CONTACTS AND LOCATIONS:
Overall Officials: Laetitia Ouedraogo Nikiema, MD, MSc, Principal Investigator — IRSS, Burkina Faso; Dominique Roberfroid, MD MSc MPhil, Study Director — ITM; Patrick Kolsteren, MD, PhD, Study Chair — ITM, Antwerpen
Locations (1):
- 18 Health Centres in Houndé District, Houndé, Burkina Faso

REFERENCES:
- [Derived] Nikiema L, Huybregts L, Kolsteren P, Lanou H, Tiendrebeogo S, Bouckaert K, Kouanda S, Sondo B, Roberfroid D. Treating moderate acute malnutrition in first-line health services: an effectiveness cluster-randomized trial in Burkina Faso. Am J Clin Nutr. 2014 Jul;100(1):241-9. doi: 10.3945/ajcn.113.072538. Epub 2014 May 7. PMID 24808482